CLINICAL TRIAL: NCT00642148
Title: A 12-week, Randomised, Double-blind, Placebo-controlled Study to Assess the Anti-inflammatory Activity, Efficacy and Safety of GW856553 in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A 12 Week Study To Assess Efficacy And Safety Of GW856553 In Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MKI102428
Record Dates: First submitted 2008-03-17; First posted 2008-03-24 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: GW856553; p38 MAPK; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — 6-(5-((cyclopropylamino)carbonyl)-3-fluoro-2-methylphenyl)-N-(2,2-dimethylprpyl)-3-pyridinecarboxamide; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Seretide (Active Comparator)
  Interventions: Drug: Placebo; Drug: Seretide
- Placebo (Placebo Comparator): Placebo tablet
  Interventions: Drug: Placebo
- GW856553 (Experimental)
  Interventions: Drug: GW856553; Drug: Placebo

INTERVENTIONS:
Drug: GW856553 — Active tablet
  Arms: GW856553
Drug: Placebo — Placebo tablet and inhaler
Drug: Seretide — Active comparator inhaler
  Arms: Seretide

SUMMARY:
Phase IIa, randomised, double-blind, double-dummy, parallel group, multi-centre study in subjects diagnosed with moderate chronic obstructive pulmonary disease (COPD). The primary objective is to evaluate the effects of 12-weeks of treatment with GW856553 7.5 mg twice daily (BID) compared with placebo on the percentage of sputum neutrophils at 12 weeks. Twelve weeks of treatment with SERETIDE 50/500 BID will be compared with placebo for effect on sputum neutrophils as a positive control arm in the study

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible for enrolment in the study must meet all of the following criteria:

* Male adults or female adults of non-childbearing potential who are between 40 and 75 years of age (inclusive). Note: a female is eligible to enter and participate in the study if she is of non-childbearing potential (i.e. physiologically incapable of becoming pregnant). This includes any female who is post-menopausal. For the purposes of this study, post menopausal is defined as being amenorrhoeic for greater than 1 year with an appropriate clinical profile, e.g. age appropriate, history of vasomotor symptoms. Postmenopausal status may be confirmed by serum FSH and oestradiol concentrations at screening if deemed necessary by the PI. Surgical sterility will be defined as females who have had a hysterectomy and/or bilateral oophorectomy or tubal ligation.
* Chronic obstructive pulmonary disease diagnosis: an established clinical history of COPD in accordance with the following description by the American Thoracic Society/European Respiratory Society [American Thoracic Society / European Respiratory Society, 2004] Chronic obstructive pulmonary disease is a preventable and treatable disease characterised by airflow limitation that is not fully reversible. The airflow limitation is usually progressive and is associated with an abnormal inflammatory response of the lungs to noxious particles or gases, primarily caused by cigarette smoking. Although COPD affects the lungs, it also produces significant systemic consequences.
* Subjects with a cigarette smoking history of ≥10 pack years (1 pack year = 20 cigarettes smoked per day for 1 year or the equivalent). Both current and former smokers are eligible to be enrolled. A former smoker is defined as a subject who has not smoked for ≥6 months at Visit 1.
* Subjects with a post-bronchodilator FEV1 to FVC ratio (FEV1:FVC) < 0.7 at Visit 1. Subjects will be assessed 30 (± 5) minutes after receiving salbutamol 400 μg.
* Subjects with a post-bronchodilator FEV1 ≥ 50% and < 80% of predicted normal for height, age and sex at Visit 1. Subjects will be assessed 30 (± 5) minutes after receiving salbutamol 400 μg.
* Subjects capable of providing signed written informed consent to participate.
* Subjects must have a QTc <450 msec on baseline ECG or triplicate ECG averaged over a brief recording interval. For subjects with baseline bundle branch block the QTc will be <480msec on baseline ECG or triplicate ECG averaged over a brief recording interval.
* A subject will be eligible for randomisation at the end of the run-in period only if the following additional criterion applies: Subjects with no evidence of an ongoing acute infection or sinus symptoms Specific information regarding warnings, precautions, contraindications, AEs, and other pertinent information on the investigational product that may impact subject eligibility is provided in the Investigator Brochure/Investigator Brochure supplement(s), product label, and other pertinent documents.

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

* Women who are pre-menopausal and of child-bearing potential, or pregnant.
* Subjects with a primary diagnosis of asthma or α-1 antitrypsin deficiency.
* Subjects who have required hospitalisation or treatment with oral corticosteroids and/or antibiotic therapy for acute worsening of COPD or lower respiratory tract infection in the 6 weeks prior to Visit 1
* Subjects with active tuberculosis or being treated for active tuberculosis, sarcoidosis or clinically overt bronchiectasis.
* Subjects with a history of any type of malignancy with the exception of successfully treated squamous cell cancer of the skin.
* Subjects with rheumatoid arthritis, connective tissue disorders and other conditions known to be associated with chronic inflammation (e.g. inflammatory bowel disease).
* Subjects with chronic infections such as gingivitis, periodontitis, prostatitis, gastritis, and urinary tract infections.
* Subjects with any acute infection, sinus symptoms, or significant trauma (burns, fractures).
* Subjects with clinically significant renal disease, diabetes mellitus/metabolic syndrome, hypertension or any other clinically significant cardiovascular, neurological, endocrine, or haematological abnormalities that are uncontrolled on permitted therapy (see Section 6.6.1).
* Subjects with clinically significant gastrointestinal or hepatic abnormalities.
* Subjects with hypoxaemia. (All subjects must have an O2 saturation of ≥ 88% on room air).
* History of Gilbert's syndrome. Subjects with a total bilirubin concentration above the upper limit of normal at Visit 1 will be excluded.
* Liver function tests (bilirubin, ALT, or AST) above upper limit of normal at Visit 1. The subject has a positive Hepatitis B surface antigen or Hepatitis C antibody result within 3 months of the start of the study.The subject has a history of HIV or other immunosuppressive disease.
* Subjects who have undergone recent surgery including lung volume reduction surgery or have conditions that prevent them from performing spirometry.
* Subjects with a history (or suspected history) of alcohol misuse or any other substance abuse.
* The subject has a three month prior history of regular alcohol consumption exceeding an average weekly intake of > 21 units (or an average daily intake of greater than 3 units) for males, or an average weekly intake of > 14 units (or an average daily intake of greater than 2 units) for females. 1 unit is equivalent to a half-pint (284mL) of beer/lager; 25mL measure of spirits or 125mL of wine; or a positive alcohol breath test at the screening visit
* Subjects who will commence or who are likely to commence statin therapy (3-hydroxy-3-methylglutaryl coenzyme A reductase inhibitors) or treatment with intranasal or topical corticosteroids, acetylsalicyclic acid, non-steroidal anti-inflammatory drugs, gemfibrozil, clopidogrel, abciximab, peroxidase proliferator-activated receptor γ agonists (e.g, rosiglitazone), fibrates, or niacin from Visit 1 until study completion. (Subjects who are receiving these medications at a stable dose at Visit 1 may be entered in the study.)
* Subjects who require treatment with any of the following from the Visit 1 until study completion:

  * Inhaled corticosteroids
  * Inhaled cromolyn sodium or nedocromil
  * Xanthines (theophylline preparations)
  * Leukotriene modifiers
  * Tiotropium
  * Long-acting inhaled β2-agonists (salmeterol, formoterol)
  * Oral β2-agonists
  * Macrolide antibiotics for more than five days
* Subjects who have received treatment with oral, intravenous or intra-articular corticosteroids within 6 weeks of Visit 1 or thereafter.
* Subjects with any known hypersensitivity to salbutamol or ipratropium bromide.
* Subjects who are participating or plan to participate in the active phase of a pulmonary rehabilitation programme during the study. Maintenance rehabilitation is permitted.
* Subjects who have received an investigational drug within 30 days or within five drug half-lives of the investigational drug (whichever is longer).
* Subjects with any clinically relevant abnormality detected by the assessments at Visit 1
* An unwillingness of male subjects to abstain from sexual intercourse with pregnant or lactating women; or unwillingness of the male subject to use a condom/spermicide in addition to having their female partner use another form of contraception such as an intra-uterine devices, diaphragm with spermicide, oral contraceptives, injectable progesterone, subdermal implants or a tubal ligation if the woman could become pregnant from the time of the first dose of investigational product for the duration of the study (i.e., through the follow-up phase).
* Subjects who have had a close household contact treated for active tuberculosis within the past 12 months, or who in the judgement of the investigator are at high risk for developing active tuberculosis, shall be excluded from the study.
* A subject will not be eligible for randomisation at the end of the run-in period if either of the following criteria applies:

  * Subjects who have experienced an exacerbation during the run-in period requiring treatment with oral corticosteroids and/or antibiotics and/or hospitalisation.
  * Subjects who are unable to produce an induced sputum sample.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2008-02-14 (Actual); Primary Completion 2009-07-27 (Actual); Study Completion 2009-07-27 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in percentage of neutrophils in induced sputum at Week 12 | Baseline (Week 0) and Week 12
  Induced sputum samples were collected at Baseline (Week 0), Week 4 and at Week 12 to evaluate the effects of 12 weeks of treatment with GW856553 7.5 mg twice daily. Baseline was defined at Week 0. Change from Baseline in neutrophil count was calculated as the Week 12 value minus the Baseline value (percentage of neutrophil of total cells in induced sputum at Week 12 minus the Baseline value). Data for adjusted mean was presented for least square mean.

SECONDARY OUTCOMES:
Change from Baseline in Plethysmography measures at Week 12 | Baseline (Week 0) and Week 12
  Plethysmography was performed to assess inspiratory capacity (IC), residual volume (RV), thoracic gas volume (TGV) at Functional Residual Capacity, Total Lung Capacity (TLC) and Slow Vital Capacity (SVC) at baseline and up to Week 12. Baseline was defined at Week 0. Change from Baseline in Plethysmography was calculated as the Week 12 value minus the Baseline value. Data for adjusted mean was presented for least square mean.
Change from Baseline in pulmonary function assessed by forced vital capacity (FVC), forced expiratory volume in 1 second (FEV1) at Week 12 | Baseline (Week 0) and Week 12
  Pre and post bronchodilator FVC and FEV1 values were calculated to assess the pulmonary function. FVC was defined as the total amount of air exhaled during the lung function test and FEV1 was defined as the amount of air which was forcibly exhaled from the lungs in the first second of a forced exhalation. Baseline was defined at Week 0. Change from Baseline in pulmonary function was calculated as the Week 12 value minus the Baseline value. Data for adjusted mean was presented for least square mean.
Change from Baseline in pulmonary function assessed by FEV1/FVC at Week 12 | Baseline (Week 0) and Week 12
  Pre and post bronchodilator FEV1/FVC ratio was measured at baseline and up to Week 12. Baseline was defined at Week 0. Change from Baseline in FEV1/FVC ratio was calculated as the Week 12 value minus the Baseline value.
Change from Baseline in pulmonary function assessed by impulse oscillometry [Peripheral airway resistance (R5 - R15)] at Week 12 | Baseline (Week 0) and Week 12
  Pulmonary function was assessed by impulse oscillometry for pre and post bronchodilator peripheral airway resistance (R5 - R15) at Baseline and up to Week 12. Baseline was defined at Week 0. Change from Baseline in pulmonary function was calculated as the Week 12 value minus the Baseline value. Data for adjusted mean was presented for least square mean.
Change from Baseline in pulmonary function assessed by impulse oscillometry: Total resistance (R5) and large airway resistance (R25) of the lung at Week 12 | Baseline (Week 0) and Week 12
  Pulmonary function was assessed by impulse oscillometry for pre and post bronchodilator Total resistance (R5) and large airway resistance (R25) at Baseline and up to Week 12. Baseline was defined at Week 0. Change from Baseline in pulmonary function was calculated as the Week 12 value minus the Baseline value.
Change from Baseline in pulmonary function assessed by impulse oscillometry: Resonant frequency (RF) and X5 as indicators of the reactive capacitance properties of the lung at Week 12 | Baseline (Week 0) and Week 12
  Pulmonary function was assessed by impulse oscillometry for pre and post bronchodilator RF and X5 as indicators of the reactive capacitance properties of the lung at Baseline and up to Week 12. Baseline was defined at Week 0. Change from Baseline in pulmonary function was calculated as the Week 12 value minus the Baseline value.
Ratio of pulmonary function assessed by impulse oscillometry at Week 12 to Baseline: low-frequency reactance area (AX) as indicator of the reactive capacitance properties of the lung | Baseline (Week 0) and Week 12
  Pulmonary function was assessed by impulse oscillometry for pre and post bronchodilator AX as indicator of the reactive capacitance properties of the lung at Baseline and up to Week 12.
Ratio of plasma fibrinogen assessment at Week 12 to Baseline | Baseline (Week 0) and Week 12
  Blood samples for measurement of fibrinogen was collected at Baseline and up to Week 12. Data for Week 12 plasma fibrinogen assessment was reported.
Ratio of biomarker assessment: Serum Surfactant Protein D (SP-D) and Clara cell protein 16 (CCP-16) at Week 12 to Baseline | Baseline (Week 0) and Week 12
  Blood samples for assessment of systemic biomarkers i.e. SP-D and CCP-16 were collected at Baseline and Up to Week 12. Ratio of geometric means at Week 12 to Baseline has been presented.
Ratio of High Sensitivity C-reactive Protein (hsCRP) at Week 12 to Baseline | Baseline (Week 0) and Week 12
  Blood samples for assessment of systemic biomarker i.e. hsCRP were collected at Baseline and Up to Week 12. Ratio of geometric means at Week 12 to Baseline has been presented.
Ratio of biomarker assessment: Interleukin 6 (IL-6), Interleukin 8 (IL-8) Matrix Metallopeptidase 9 (MMP-9) and PARC (Pulmonary and activation-regulated chemokine) at Week 12 to Baseline | Baseline (Week 0) and Week 12
  Blood samples for assessment of systemic biomarkers i.e. IL-6, IL-8, MMP-9 and PARC were collected at Baseline and Up to Week 12. Adjusted ratio to Baseline value at Week 12 has been presented.
Ratio of biomarker sorbitol-Induced phosphorylated heat shock protein (pHSP-27) in whole blood pre-dose and 2 h post-dose assessment at Week 12 to Baseline | Baseline (Week 0) and Week 12
  Levels of ex vivo pHSP27 in whole blood pre-dose and 2 hours post-dose at selected centres was assessed over 12 Weeks of treatment. Adjusted ratio to Baseline value at Week 12 has been presented.
Ratio of biomarker LPS-Induced TNFα Release (pre and post dose) assessment at Week 12 to Baseline | Baseline (Week 0) and Week 12
  Levels of ex vivo LPS induced TNF-a in whole blood pre-dose and 2 hours post-dose at selected centres was assessed over 12 Weeks of treatment. Adjusted ratio to Baseline value at Week 12 has been presented.
Ratio of total leukocyte count in induced sputum assessments at Week 12 to Baseline | Baseline (Week 0) and Week 12
  Induced sputum samples for assessment of total cell count were collected at Baseline (Week 0), Week 4 and at Week 12 to evaluate the effects of 12 weeks of treatment with GW856553 7.5 mg twice daily. Adjusted ratio to Baseline value at Week 12 has been presented.
Change from Baseline in sputum assessment for macrophages as a percentage of total cells at Week 12 | Baseline (Week 0) and Week 12
  Percentage of total cells for macrophages was assessed in induced sputum at Baseline and up to Week 12. Baseline was defined at Week 0. Change from Baseline in Percentage of total cells for macrophages was calculated as the Week 12 value minus the Baseline value. Data for adjusted mean was presented for least square mean.
Change from Baseline in sputum assessment for lymphocytes and eosinophils as a percentage of total cells at Week 12 | Baseline (Week 0) and Week 12
  Percentage of total cells for lymphocyte and eosinophil was assessed in induced sputum at Baseline and up to Week 12. Baseline was defined at Week 0. Change from Baseline in Percentage of total cells for macrophages was calculated as the Week 12 value minus the Baseline value.
Change from Baseline in sputum assessment for lymphocytes and eosinophils as absolute inflammatory cell numbers at Week 12 | Baseline (Week 0) and Week 12
  Absolute inflammatory cell numbers for lymphocyte and eosinophil was assessed in induced sputum at Baseline and up to Week 12. Baseline was defined at Week 0. Change from Baseline in Absolute inflammatory cell numbers for lymphocyte and eosinophil was calculated as the Week 12 value minus the Baseline value.
Ratio of sputum assessment for Neutrophils and macrophages as absolute inflammatory cell numbers at Week 12 to Baseline | Baseline (Week 0) and Week 12
  Absolute inflammatory cell numbers for neutrophils and macrophages was assessed in induced sputum at Baseline and up to Week 12. Adjusted ratio to Baseline value at Week 12 has been presented.
Ratio of sputum weight and volume at Week 12 to Baseline | Baseline (Week 0) and Week 12
  Induced sputum weight and volume was assessed up to Week 12. For participants who were not able to produce an induced sputum sample after induction (and for these participants only), missing values were imputed with half lowest weight. Adjusted ratio to Baseline value at Week 12 has been presented.
Ratio of concentration of inflammatory biomarkers (ng/ml)-myeloperoxidase (MPO) at Week 12 to Baseline | Baseline (Week 0) and Week 12
  Sputum samples were analyzed to determine the concentration of inflammatory biomarker i.e MPO up to Week 12. Adjusted ratio to Baseline value at Week 12 has been presented.
Ratio of concentration of inflammatory biomarkers (ug/ml)- total protein at Week 12 to Baseline | Baseline (Week 0) and Week 12
  Sputum samples were analyzed to determine the concentration of inflammatory biomarker i.e total protein up to Week 12. Adjusted ratio to Baseline value at Week 12 has been presented.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (28):
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- GSK Investigational Site, Helsinki, Finland
- Germany (6):
  - GSK Investigational Site, Gauting, Bavaria
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Großhansdorf, Schleswig-Holstein
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Berlin
- GSK Investigational Site, Riga, Latvia
- GSK Investigational Site, Klaipėda, Lithuania
- Netherlands (3):
  - GSK Investigational Site, Breda
  - GSK Investigational Site, Heerlen
  - GSK Investigational Site, Veldhoven
- New Zealand (2):
  - GSK Investigational Site, Auckland
  - GSK Investigational Site, Wellington
- Russia (3):
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
- Slovenia (2):
  - GSK Investigational Site, Kamnik
  - GSK Investigational Site, Ljubljana
- South Africa (3):
  - GSK Investigational Site, Cape Town, Gauteng
  - GSK Investigational Site, eManzimtoti
  - GSK Investigational Site, Mowbray
- GSK Investigational Site, Seoul, South Korea
- United Kingdom (3):
  - GSK Investigational Site, Headington, Oxfordshire
  - GSK Investigational Site, Cottingham, East Yorkshire
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Lomas DA, Lipson DA, Miller BE, Willits L, Keene O, Barnacle H, Barnes NC, Tal-Singer R; Losmapimod Study Investigators. An oral inhibitor of p38 MAP kinase reduces plasma fibrinogen in patients with chronic obstructive pulmonary disease. J Clin Pharmacol. 2012 Mar;52(3):416-24. doi: 10.1177/0091270010397050. Epub 2011 Nov 16. PMID 22090363
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: MKI102428 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: MKI102428 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: MKI102428 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: MKI102428 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: MKI102428 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: MKI102428 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: MKI102428 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register